CLINICAL TRIAL: NCT05863455
Title: Effect of Mild Sedation and Analgesia on Radial Artery Cannulation in Novice Residents: a Prospective, Randomized Controlled Trial
Brief Title: Effect of Mild Sedation and Analgesia on Radial Artery Cannulation in Novice Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Principal investigator, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-KY-297
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Sedation and Analgesia
Keywords: Radial Artery Cannulation; Novice Operators
MeSH Terms: conditions — Agnosia | interventions — Analgesia; Sufentanil; Midazolam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mild sedation and analgesia (Experimental): Intravenous injection of 0.1ug/kg sufentanil and 0.03mg/kg midazolam for sedation and analgesia before radial artery cannulation.
  Interventions: Drug: mild sedation and analgesia
- control (Active Comparator): Intravenous injection of an equivalent volume of saline before radial artery cannulation.
  Interventions: Drug: control

INTERVENTIONS:
Drug: mild sedation and analgesia — Intravenous injection of 0.1ug/kg sufentanil and 0.03mg/kg midazolam for sedation and analgesia before radial artery cannulation
  Other Names: sufentanil and midazolam
  Arms: mild sedation and analgesia
Drug: control — ntravenous injection of an equivalent volume of saline before radial artery cannulation.
  Other Names: saline
  Arms: control

SUMMARY:
The aim of this study is to conduct a prospective, single-center randomized controlled study to investigate the effect of mild midazolam combined with sufentanil on radial artery cannulation in novice operators.

DETAILED DESCRIPTION:
outcome: patients discomfort，visual analogue scale，First-attempt success rate，the success rate of radial artery cannulation within 10 minutes, Complication rate

ELIGIBILITY:
Inclusion Criteria:

* Patients who required arterial cannulation for continuous blood pressure monitoring
* Aged >20years
* ASA physical status of 1-3
* BMI 18-28kg/m2
* All patients agreed to participate in this study at the time of recruitment and signed an informed consent form.

Exclusion Criteria:

* a positive Allen's test
* infection at the puncture site
* coagulation disorders; arterial diseases (such as Raynaud's disease or thromboangiitis obliterans)
* use of vasoactive drugs within 30 minutes before measurement during the study
* patients with arterial abnormalities and bends; hemorrhagic shock
* arterial atherosclerosis; radial artery puncture within the past 30 days
* chronic use of opioid or benzodiazepine drugs
* and known allergies or adverse reactions to benzodiazepines or opioids.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Overall success rate | During radial artery cannulation (up to 1 hour)
  success rate of puncture and catheter placement within 10 minutes.

SECONDARY OUTCOMES:
patients discomfort | During radial artery cannulation (up to 1 hour)
  0 corresponding to "no anxious", 1 corresponding to "mildly anxious", 2 corresponding to "moderately anxious" and 3 corresponding to "very anxious"
visual analogue scale | During radial artery cannulation (up to 1 hour)
  ranging from 0 to 10 was emplyed to assess pain intensity
First-attempt success rate | During radial artery cannulation (up to 1 hour)
  Success at the first skin puncture
Complication rate | postoperative 1 day and 3 day
  Hematoma, Distal ischemia, Spasm accessed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Qinghe Zhou, Principal Investigator — Affiliated Hospital of Jiaxing University
Locations (1):
- Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xi YZ, Li ZP, Zhou QH. Effect of mild sedation and analgesia on radial artery cannulation in novice residents: a prospective, randomized controlled trial. BMC Med Educ. 2024 Dec 21;24(1):1515. doi: 10.1186/s12909-024-06568-8. PMID 39709419